CLINICAL TRIAL: NCT05296122
Title: Safety and Feasibility of MR-guided Laser Thermal Ablation of Brain Lesion Using the Tranberg® Thermal Therapy System and Tranberg® Thermoguide Workstation
Brief Title: Safety and Feasibility of MR-guided Laser Thermal Ablation of Brain Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Laserthermia Systems AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CTP-2021-012
Record Dates: First submitted 2022-02-15; First posted 2022-03-25 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Glioblastoma
Keywords: Laser Thermotherapy; Magnetic Resonance guidance; Interventional; Thermal ablation; Clearpoint Neuro Navigation; Magnetic Resonance thermometry; Minimal invasive; MRg LITT; TRANBERG; Thermoguide; Stereotactic Laser Ablation
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): MR-Guided Laser Thermal ablation of brain lesions using the TRANBERG® Thermal Therapy System and TRANBERG ® Thermoguide Workstation.
  Interventions: Device: TRANBERG® laser applicators when used in MR-guided laser thermal ablation of brain lesions using the TRANBERG® Thermal Therapy System and TRANBERG® Thermoguide Workstation.

INTERVENTIONS:
Device: TRANBERG® laser applicators when used in MR-guided laser thermal ablation of brain lesions using the TRANBERG® Thermal Therapy System and TRANBERG® Thermoguide Workstation. — The main purpose with the study is to investigate safety and feasibility of the TRANBERG® laser applicators when used in MR-guided laser thermal ablation of brain lesions using the TRANBERG® Thermal Therapy System and TRANBERG® Thermoguide Workstation together with SmartTwist™ MR Hand Drill with the SmartTip™ MR Drill Kit for MR-guided laser thermal ablation of brain lesions.

SUMMARY:
This will be an open-label, pilot, exploratory, single centre clinical investigation. This is an early feasibility single arm study. No formal hypothesis is proposed. A total of up to 15 evaluable subjects receiving a non-radical ablation is planned.

The safety and feasibility outcomes will be measured directly post-treatment, 48h and 3 months post-treatment.

A minimal invasive neurosurgical approach with a Magnetic Resonance Imaging (MRI)-based stereotactic guidance system will be utilized for the planning, navigation, intracranial access, placement and confirmation of the Laser applicator prior to ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Lesions eligible for Laser Interstitial ThermoTherapy (LITT), target tumor ≤10cc in volume
2. Age ≥ 18 and < 80 years
3. Ability to undergo contrast-enhanced Computed Tomography (CT), Positron Emission Tomography (PET)-CT and contrast-enhanced MRI.
4. Women of childbearing potential must have a negative pregnancy test.
5. Eastern Cooperative Oncology Group (ECOG) performance status of ≤2
6. Primary glioblastoma/astrocytoma WHO grade IV confirmed by 1)Magnetic Resonance Imaging according to RANO citera and 2)Frozen section biosy diagnosis, and considered not suitable for open surgery or other primary treatment, or Recurrent glioblastoma/astrocytoma WHO grade IV confirmed by Magnetic Resonance Imaging according to RANO criteria.
7. ≥3 months since last radiotherapy of the brain
8. Supratentorial tumor localization with or without prior surgery for recurrence.
9. Life expectancy of ≥3 months
10. The subject reports having understood and has signed the Informed Consent Form (ICF) and is willing to comply with all investigation visits and assessments.
11. Anticipated compliance with treatment and follow-up

Exclusion Criteria:

1. Subject contraindicated for MRI, including subjects who may have contraindications due to implanted medical devices
2. Subject evaluated not to be fit for surgery due to liver/kidney/other organ dysfunction verified by laboratory tests
3. Identified intratumoral cystic or haemorrhagic transformation in target tumor
4. Known bleeding disorder
5. ECOG performance status of >2
6. Previous (within 30 days prior to enrollment / randomization) and concurrent treatment during the treatment phase with other investigational drug/s or device/s
7. Pregnancy or breastfeeding
8. The subject has a cognitive incapacity or language barrier precluding adequate understanding or cooperation
9. The subject is considered by the Investigator to be unsuitable to participate in the investigation for any other reason.
10. Any severe diseases interfering with the performance, evaluation, and outcome of the clinical evaluation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Device and procedure related adverse events | From Day 1 throughout the study until 3 months
  The number and severity of adverse events related to the TRANBERG® Laser applicator when used in MR-guided laser thermal ablation of brain lesions

SECONDARY OUTCOMES:
Device and procedure related adverse events | From Day 1 throughout the study until 3 months
  The number and severity of adverse events related to the SmartTwist™ MR HAND DRILL with the SmartTip™ MR Drill Kit when used for intracranial access.

OTHER OUTCOMES:
Device performance | At 3 months after treatment
  The volume of remaining tumor mass will be assessed by contrast enhanced MRI after MR-Guided laser thermal ablation using the TRANBERG® Thermal Therapy System and TRANBERG® Thermoguide Workstation.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Siesjö, Prof, Principal Investigator — Department of Neurosurgery, Skåne University Hospital, 22185 Lund,Sweden
Locations (1):
- Department of Neurosurgery, Skåne University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No